CLINICAL TRIAL: NCT07377955
Title: Combined Volume Guarantee High-Frequency Oscillatory Ventilation (HFOV-VG) Versus Conventional High-Frequency Oscillatory Ventilation (HFOV) on Grade 2 to 3 Bronchopulmonary Dysplasia (BPD) or Death in Preterm Infants <32 Weeks With Respiratory Distress Syndrome (RDS)
Brief Title: Combined Oscillation-Volume guarantEe Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xingwang Zhu (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); The Affiliated Hospital of Jining Medical University and Zaozhuang City (Unknown); Chongqing Qianjiang Central Hospital (Unknown); First People's Hospital of Chenzhou (Other); Fujian Children's Hospital (Unknown); Fuling Hospital of Chongqing University (Unknown); Guangdong Women and Children Hospital (Other); Henan Children's Hospital Zhengzhou Children's Hospital (Unknown); Hunan Children's Hospital (Other Government); Hunan Provincial Maternal and Child Health Care Hospital (Other); Hunan Provincial People's Hospital (Other); Inner Mongolia Maternal and Child Health Care Hospital (Other); Jiangxi Maternal and Child Health Hospital (Other); Kunming Children's Hospital (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Moscow Regional Research Institute of Obstetrics and Gynecology named after Academician V. I. Krasnopolsky (Unknown); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); People's Hospital of MeiShan (Unknown); Quanzhou Women's and Children's Hospital (Unknown); Qujing Maternal and Child Hospital (Unknown); Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University (Unknown); Shandong Provincial Maternal and Child Health Care Hospital Affiliated to Qingdao University (Unknown); Shanxi Women and Children Hospital (Unknown); Shenzhen Longhua Maternity and Child Health Care Hospital (Unknown); Shijiazhuang Obstetrics and and Gynecology Hospital (Unknown); Third Affiliated Hospital of Guangzhou Medical University (Unknown); Women and Children's Hospital of Chongqing Medical University (Unknown); Women and Children's Hospital of Ningbo University (Unknown); Zhangzhou Affiliated Hospital of Fujian Medical School (Unknown)
Responsible Party: Sponsor-Investigator, Xingwang Zhu, Director, Jiulongpo No.1 People's Hospital
Organization: Jiulongpo No.1 People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Combined Oscillation-Volume gu
Record Dates: First submitted 2026-01-15; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Distress Syndrome (& [Hyaline Membrane Disease]); Bronchopulmonary Dysplasia (BPD)
MeSH Terms: conditions — Respiratory Distress Syndrome; Hyaline Membrane Disease; Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFOV (Active Comparator): HFOV: 1) Mean airway pressure (MAP) and FiO2: titrated via oxygenation-guided lung recruitment maneuvers21-23 to maintain preductal SpO2 target of 89%-94%. 2) Frequency: 12-15 Hz for birth weight (BW)<1500g, and 10-12 Hz for BW≥ 1500g. 3) I:E ratio: 1:1 or 1:2 according to recommendations of manufacturers and local habits
  Interventions: Device: HFOV
- HFOV+VG (Active Comparator): HFOV-VG Group: ①VThf: <1000g 1.5-1.8ml/kg, 1000-1500g 1.8-2.2ml/kg, >1500g, 2.2-2.5ml/kg; ②Amplitude automatically adjusted by volume guarantee algorithm and the upper limit was set at 15% above the measured value after achieving the target VThf, with the constraint that it must not exceed 20 cm H2O for BW<1000g, 25cm H2O for BW 1000-1500g or 25-30 cmH2O for BW>1500g; ③If the target VThf is not achieved after the amplitude has reached its upper limit, airway issues (e.g., suctioning) or lung recruitment should be addressed first, rather than overriding the amplitude limit.
  Interventions: Device: HFOV+VG

INTERVENTIONS:
Device: HFOV — HFOV: 1) Mean airway pressure (MAP) and FiO2: titrated via oxygenation-guided lung recruitment maneuvers to maintain preductal SpO2 target of 89%-94%. 2) Frequency: 12-15 Hz for birth weight (BW)<1500g, and 10-12 Hz for BW≥ 1500g. 3) I:E ratio: 1:1 or 1:2 according to recommendations of manufacturers and local habits
  Arms: HFOV
Device: HFOV+VG — HFOV-VG Group: ①VThf: <1000g 1.5-1.8ml/kg, 1000-1500g 1.8-2.2ml/kg, >1500g, 2.2-2.5ml/kg; ②Amplitude automatically adjusted by volume guarantee algorithm and the upper limit was set at 15% above the measured value after achieving the target VThf, with the constraint that it must not exceed 20 cm H2O for BW<1000g, 25cm H2O for BW 1000-1500g or 25-30 cmH2O for BW>1500g; ③If the target VThf is not achieved after the amplitude has reached its upper limit, airway issues (e.g., suctioning) or lung recruitment should be addressed first, rather than overriding the amplitude limit
  Arms: HFOV+VG

SUMMARY:
Respiratory Distress Syndrome (RDS) remains the most common respiratory complication in the early postnatal period among preterm infants born before 32 weeks' gestational age. For this population, implementing lung-protective ventilation strategies is essential to shorten the duration of intubation, reduce the incidence and severity of bronchopulmonary dysplasia (BPD), lower mortality, and improve overall outcomes.

HFOV-VG was first reported in 2015 to be safely applied in neonates. The fundamental principle lies in its ability to stabilize the tidal volume of high-frequency ventilation (VThf), thereby reducing sheer stress from amplitude fluctuations, while simultaneously permitting lower VThf settings to minimize volutrauma.

This study aims to evaluate whether HFOV+VG is superior to HFOV in reducing the composite outcome of grade 2-3 BPD or death at 36 weeks' post-menstrual age (PMA).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 24+0/7< 320/7 weeks
* Diagnosis of RDS within 72 hours after birth, requiring endotracheal ventilation for both elective and rescue HFOV

Exclusion Criteria:

* Severe birth defects: severe congenital heart disease, diaphragmatic hernia, gastrointestinal malformations, congenital brain developmental abnormalities, congenital pulmonary cysts
* Uncorrected shock
* Existence of grade 3-4 IVH before ventilated
* Other conditions deemed unsuitable for enrollment by neonatologists, including endotracheal intubation performed specifically for the purpose of the INSURE or INRECSURE technique.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of grade 2-3 BPD or in-hospital death at 36 weeks' PMA | 36 weeks gestational age

SECONDARY OUTCOMES:
In-hospital death at 36 weeks' PMA | 36 weeks gestational age
The incidence of BPD at 36 weeks' PMA | 36 weeks gestational age
The duration of invasive ventilation at the time of the first successful extubation | through study completion, an average of 1 year
Surfactant doses | through study completion, an average of 1 year
The incidence of normocapnia, hypercapnia, and hypocapnia during the intervention period | through study completion, an average of 1 year
Pulmonary hypertension (PH) requiring iNO treatment, including PPHN within 7 days after birth and cPH after 28 days of life | through study completion, an average of 1 year
hsPDA (Iowa score ≥6 ) | through study completion, an average of 1 year
The incidence of massive pulmonary hemorrhage, pneumothorax, pneumomediastinum, pneumopericardium, and ventilator-associated pneumonia(VAP) | through study completion, an average of 1 year
The incidence of Grade III to IV IVH according to Papile 1978 criteria | through study completion, an average of 1 year
The incidence of Necrotizing enterocolitis (NEC) > grade II according to Modified Bell's Staging Criteria | through study completion, an average of 1 year
The incidence of Culture-proven late-onset sepsis (onset after 72 hours of life) | through study completion, an average of 1 year
The incidence of Retinopathy of premature > grade II | through study completion, an average of 1 year
The duration of hospitalization | through study completion, an average of 1 year
Weight gain (g/kg/day) | through study completion, an average of 1 year
The incidence of discharge against medical advice (DAMA) | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Yes
Researchers who wish to use the data may apply by emailing the principal investigator with a comprehensive study protocol. After the primary results of this trial have been published, the full, de-identified dataset will be made available to all participating sites of COVES for secondary analyses.
Supporting Information: Study Protocol, SAP